CLINICAL TRIAL: NCT00549055
Title: A Study On The Efficacy Of Macugen Injections In Patients With Neovascular Age-Related Macular Degeneration (AMD) In Real Life (Macureli Study).
Brief Title: A Study On The Efficacy Of Macugen Injections In Patients With Neovascular Age-Related Macular Degeneration In Real Life.
Acronym: MACURELI
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751026
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Macugen Age-related macular degeneration (AMD) Observational study
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who obtained reimbursement of Macugen.
  Interventions: Drug: Macugen

INTERVENTIONS:
Drug: Macugen — Dosage form: solution for injection (intravitreal) Dosage: 0.3mg Frequency: every 6 weeks (9 injections/year)
  Other Names: Pegaptanib sodium

SUMMARY:
To assess effectiveness of Macugen for treatment of neovascular age-related macular degeneration by measuring the evolution of visual acuity. Treatment duration, frequency of administration and combination with other treatments will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with subfoveal neovascular (wet) age-related macular degeneration
* Patients having received at least 1 Macugen injection
* Treatment naive patients, or patients having received conventional therapy
* Patients having signed and dated informed consent.

Exclusion Criteria:

* Patients participating in another clinical study with Macugen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who obtained reimbursement for Macugen, recruited by retina specialists from ophthalmology centres with experience in intravitreal injections.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Belgium (4):
  - Pfizer Investigational Site, Aarschot
  - Pfizer Investigational Site, Deurne
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751026&StudyName=A%20study%20on%20the%20efficacy%20of%20Macugen%20injections%20in%20Patients%20with%20Neovascular%20Age-Related%20Macular%20Degeneration%20in%20real%20life.

RESULTS

PARTICIPANT FLOW:
Groups:
- Macugen: Intraocular injections of Macugen into the treated eye. The use and dosage recommendations for Macugen took place on the basis of the approved package insert.
Period: Overall Study
Arm/Group | Macugen
Started | 38
Completed | 3
Not Completed | 35
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 18
Not completed — Stabilization | 5
Not completed — Progression to fibrosis | 2
Not completed — Decrease of size | 1
Not completed — Active choroidal neovascula increased | 1
Not completed — Vitreous hemorrhage | 1
Not completed — Growth choroidal neovascularisation | 1
Not completed — Choroidal neovascularization | 1
Not completed — Very low visual acuity (VA) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Macugen
Number analyzed (Participants) | 38
Age, Customized [Number; unit: Participants]
  < 65 years | 3
  65 to 74 years | 8
  75 to 84 years | 22
  >= 85 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Final Visit in Visual Acuity (VA) Score
Description: Best corrected VA score, assessed on the scale over time (best corrected VA score at Final Visit minus best corrected VA score at Baseline). Lower scores represent poorer eyesight and higher scores represent better eyesight with a value of 1 representing normal eyesight. A positive change in score represents an improvement in sight.
Time Frame: Baseline, Month 24 or Early Termination
Population: The Full Analysis Set (FAS) was derived from the set of all enrolled participants who were administered at least 1 injection of the study medication and had at least 1 post Baseline efficacy measurement. Participants analyzed refers to number of participants with analyzable data.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Macugen
Number analyzed (Participants) | 28
Scores on scale | -0.044 (0.122)

2. Secondary Outcome: Number of Participants With Change in VA: Improvement
Description: Investigator's clinical judgement of Improvement in status of vision as compared to the previous Macugen injection, calculated from measurement of the difference between the VA scores at the 2 visits.
Time Frame: Months 3, 6, 9 and 12
Population: FAS; n= number of participants with analyzable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 30
Participants
  Month 3 (n=18) | 3
  Month 6 (n=5) | 1
  Month 9 (n=2) | 1
  Month 12 (n=2) | 1

3. Secondary Outcome: Number of Participants With Change in VA: Stabilization
Description: Investigator's clinical judgement as Stabilization in status of visual acuity as compared to the previous Macugen injection, determined from measurement difference between the VA scores at the 2 visits.
Time Frame: Months 3, 6, 9 and 12
Population: FAS; n= number of participants with analyzable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 30
Participants
  Month 3 (n=18) | 11
  Month 6 (n=5) | 2
  Month 9 (n=2) | 0
  Month 12 (n=2) | 1

4. Secondary Outcome: Number of Participants With Change in VA: Worsening
Description: Investigator's clinical judgement as Worsening in status of vision as compared to the previous Macugen injection, determined from measurement difference between the VA scores at the 2 visits.
Time Frame: Months 3, 6, 9 and 12
Population: FAS; n= number of participants with analyzable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 30
Participants
  Month 3 (n=18) | 4
  Month 6 (n=5) | 2
  Month 9 (n=2) | 1
  Month 12 (n=2) | 0

5. Secondary Outcome: Duration of Treatment
Description: Duration of treatment per participant calculated as: date of injection (for the last injection of Macugen) minus date of injection (for the first injection of Macugen).
Time Frame: Baseline up to 28.4 months
Population: FAS
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Macugen
Number analyzed (Participants) | 30
Months | 4.66 (5.26)

6. Secondary Outcome: Frequency of Macugen Administration
Description: Average frequency of Macugen administration per participant calculated as: (number of Macugen injections administered per participant - 1)/ duration of treatment.
Time Frame: Baseline up to 28.4 months
Population: FAS
Measure: Mean (Standard Deviation); unit: Weeks per injection
Arm/Group | Macugen
Number analyzed (Participants) | 30
Weeks per injection | 7.74 (4.80)

7. Secondary Outcome: Number of Participants Who Received Other Concomitant Age Related Macular Degeneration (AMD) Treatments
Description: Derived by whether a participant took any other AMD treatments at any time (at any Study Treatment Visit).
Time Frame: Months 3, 6, 9 and 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 30
Participants | 4

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Macugen
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=38)
Myodesopsia (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.